CLINICAL TRIAL: NCT02478073
Title: Piperacillin Pharmacokinetics in Intensive Care Unit Patients Following Standard Treatment With Intermittent and Continuous Infusion
Brief Title: Piperacillin Pharmacokinetics in ICU Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Other Study IDs: AB-ICU
Record Dates: First submitted 2015-06-15; First posted 2015-06-23 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Antibiotic dosing in critically ill patients poses a challenge for clinicians due to the pharmacokinetic changes seen in this population. Piperacillin/tazobactam is often used for empirical treatment, and initial appropriate dosing is crucial for reducing mortality.

Patients in the Intensive Care Unit (ICU), treated with piperacillin/tazobactam, had their plasma concentration of piperacillin determined 1-3 times weekly. Patients received piperacillin as intermittent bolus infusion 3 times daily or as continuous infusion (this was up to the treating physician). Time above the minimal inhibitory concentration (T>MIC) estimated for each patient was evaluated against clinical breakpoint MIC for Pseudomonas aeruginosa (16 mg/L). Pharmacokinetic-pharmacodynamic (PK-PD) targets evaluated were 100% f T>MIC (free piperacillin concentration maintained above the MIC throughout the dosing interval) and 50% fT>4xMIC (free piperacillin concentration maintained at a level fourfold the MIC for at least 50% of the dosing interval).

DETAILED DESCRIPTION:
Early appropriate antimicrobial therapy is of utmost importance for reducing mortality in critically ill patients with sepsis and septic shock. Pathophysiological changes associated with the septic process, such as changes in volume of distribution (Vd), drug clearance (CL), decrease in plasma-protein concentration and organ dysfunction, lead to pharmacokinetic (PK) changes that may alter the efficacy of the antimicrobial given. As a consequence, antibiotic plasma concentrations are variable and hard to predict in these patients, which makes optimal antibiotic exposure a challenge, especially in the early phase of treatment.

Piperacillin/tazobactam is a β-lactam - β-lactamase inhibitor combination frequently used for empirical treatment in the critically ill. It is a time-dependent antibiotic where antibacterial activity is related to the time for which the free, unbound concentration of the drug is maintained above the minimal inhibitory concentration (f T>MIC). Maximizing f T>MIC both increases the therapeutic impact and reduces the risk of drug resistance development. Because of the PK changes seen in the critically ill, standard dosing of antimicrobials may result in subtherapeutic plasma-concentrations and it has been suggested that current empiric dosing recommendations for Intensive Care Unit (ICU) patients are inadequate and needs to be reconsidered.

Piperacillin/tazobactam is generally administered either as 4g/0.5g every 8 hour (h) or as 12g given continuously over 24 hours.The aim of this study is to determine if this dosing results in therapeutic plasma concentrations in septic patients. Patients treated with piperacillin/tazobactam given as intermittent bolus infusion had piperacillin plasma concentrations determined once a week. Patients treated with piperacillin/tazobactam given as continuous infusion had piperacillin plasma concentrations determined three times a week. Time above the minimal inhibitory concentration (T>MIC) estimated for each patient was evaluated against clinical breakpoint MIC for Pseudomonas aeruginosa (16 mg/L). Pharmacokinetic-pharmacodynamic (PK-PD) targets evaluated were 100% f T>MIC (free piperacillin concentration maintained above the MIC throughout the dosing interval) and 50% fT>4xMIC (free piperacillin concentration maintained at a level fourfold the MIC for at least 50% of the dosing interval).

The unbound piperacillin plasma concentrations were determined using ultra high performance liquid chromatography (UPLC). There was no intervention in the study.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis or septic shock
* Treatment with piperacillin/tazobactam

Exclusion Criteria:

* Age under 18 years
* Renal replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with sepsis or septic shock, treated with piperacillin/tazobactam in the Intensive Care Unit (ICU).
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Blood-plasma concentration of Piperacillin | A blood-test will be drawn 1-3 times weekly. Participants will be followed for the duration of piperacillin/tazobactam treatment, an expected average time of two weeks.
  Blood-plasma concentration of Piperacillin will be performed through ultra high performance liquid chromatography (UPLC). The concentrations will be compared to the clinical breakpoint MIC for Pseudomonas aeruginosa (16 mg/L).

SECONDARY OUTCOMES:
Percentage of time above the minimal inhibitory concentration (T>MIC) | A blood-test will be drawn 1-3 times weekly. Participants will be followed for the duration of piperacillin/tazobactam treatment, an expected average time of two weeks.
  The blood-plasma concentrations will be used to determine the percentage of time, within the dosing interval, that the blood-plasma concentration is at a level above the minimal inhibitory concentration (T>MIC)

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Gjedsted, MD, PhD, Principal Investigator — Aarhus University Hospital, Department of Anesthesia and Intensive Care Medicine
Locations (1):
- Aarhus Univbersity Hospital, Department of Anesthesia and Intensive Care Medicine, Aarhus N, Denmark